CLINICAL TRIAL: NCT04946591
Title: Feasibility and Impact of ICG and 4K Overlay in Laparoscopic Hepatic Surgery on Real-time Tumor Detection: A Single-centre Prospective Study
Brief Title: Feasibility and Impact of ICG and 4K Overlay in Laparoscopic Hepatic Surgery on Real-time Tumor Detection
Acronym: LiverLight
Status: Completed | Type: Observational
Sponsor: Klinikum Saarbrücken, Klinik für Allgemein-, Viszeral- und Thoraxchirurgie, Chirurgische Onkologie (Other)
Responsible Party: Principal Investigator, Dr.med Dr. habil Gregor A. Stavrou, Head of the Department, Klinikum Saarbrücken, Klinik für Allgemein-, Viszeral- und Thoraxchirurgie, Chirurgische Onkologie
Other Study IDs: 26/21
Record Dates: First submitted 2021-06-19; First posted 2021-07-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Hepatectomy
Keywords: Indocyanine green; Tumor localization; Bile Leak; Ultra-high-definition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, resected liver specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Achievement of tumor-free resection margin with the largest possible remnant liver parenchyma is the major challenge in hepatic surgery. Therefore, perioperative tumor detection, anatomical mapping of liver segments and also nearby structures are vital to improve the short- and long-term surgical outcomes. Over last decades, several real-time methods have been introduced for this purpose. These methods are mostly based on the utilizing of traceable dyes, which are excreted into the biliary tract. With the advances in minimal invasive surgery and video technology, indocyanine green became the most used dye in this manner. It has been demonstrated that using indocyanine green, small liver tumors can be detected, which cannot be identified using conventional intraoperative methods. Based on the literature, the reported sensitivity of tumor detection using indocyanine green is ranging between 98%-100%, while conventional methods could not reach 90% sensitivity. Posthepatectomy bile leakage, as well as in- or outflow distributions due to the potential vascular reconstructions, are some of the most common complications that can occur especially after complex liver surgeries. Beside the abovementioned advantages of indocyanine green, several researchers have also shown the feasibility of indocyanine green to identify the intraoperative bile leaks and any in- or outflow distributions. Nevertheless, laparoscopic assisted liver surgery is technically challenging, mostly because of the restricted degrees of instrument movements, camera instability, and loss of depth perception. In particular, the loss of depth perception and inaccurate object localization can lead to intraoperative complications and a long learning curve. Advances in video technology, namely 4K ultra-high-definition imaging have been developed to reduce perioperative complications and to shorten the learning curve during laparoscopic liver surgery. This is the first prospective study evaluating the impact of indocyanine green imaging during 4K laparoscopic liver surgery on real-time tumor detection and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Aged above 18 years
* Undergoing any type of liver resections

Exclusion Criteria:

* Unresectable liver tumors
* Known indocyanine green allergy
* Iodine allergy
* Advanced cirrhosis (Child C)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with any type of liver tumor undergoing 4K laparoscopic hepatectomy using indocyanine green
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Tumor localization | One day

SECONDARY OUTCOMES:
Remnant liver venous drainage | One day
Detection of resection plane | One day
Rate of intraoperative bile leak | One day
  Using indocyanine green and fluorescence camera
Rate of postoperative bile leak | Three months
  Based on the ISGLS criteria
Resection margin | One day
  Using fluorescence camera
Rate of morbidity | Three months
  Based on the Clavien-Dindo classification
Duration of hospital stay | Three months
Rate of mortality | Three months
  All cause death events

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Saarbrücken, Saarbrücken, Saarland, Germany